CLINICAL TRIAL: NCT06662045
Title: Study on the Association Between Iron Deficiency Anemia and Neurobehavioral Development and Cognitive Function in Children Aged 6 to 24 Months
Brief Title: Impact of Iron Deficiency Anemia on Neurobehavioral and Cognitive Development in Children Aged 6 to 24 Months
Status: Recruiting | Type: Observational
Sponsor: Pingshan District Maternal & Child Healthcare Hospital of Shenzhen (Other)
Responsible Party: Sponsor
Other Study IDs: 20230608
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Iron-Deficiency Anemia; Neurobehavioral Manifestations; Growth Disorders; Nutritional Status
MeSH Terms: conditions — Anemia, Iron-Deficiency; Neurobehavioral Manifestations; Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Iron-Deficient Group: This group consists of children diagnosed with iron-deficiency anemia.
- Control Group (Non-Anemic): This group consists of children without iron-deficiency anemia.

SUMMARY:
The goal of this observational study is to explore the relationship between iron-deficiency anemia and neurobehavioral development in children aged 6-24 months. This study focuses on children who undergo health check-ups and blood tests at pediatric health clinics in Pingshan District, Shenzhen, China.

The main questions it aims to answer are:

How does iron-deficiency anemia affect children's neurobehavioral development, including motor skills, language ability, and social behavior? How does anemia influence growth and nutrition, such as weight, height, and body mass index (BMI) in children?

Participants will:

Undergo blood tests (including hemoglobin levels, serum ferritin, and serum iron) to assess anemia status.

Be assessed using the "Neuropsychological Behavioral Development Scale for Children Aged 0-6" to measure motor, cognitive, language, and social development.

Provide general health information, such as birth history, feeding methods, and parental details, through interviews with trained surveyors.

Researchers will compare children with and without iron-deficiency anemia to determine differences in neurobehavioral outcomes and development levels. The findings aim to provide evidence for early interventions to prevent the negative impacts of anemia and support children's healthy development.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 24 months at the time of enrollment
* Diagnosed with iron-deficiency anemia (for the exposure group) or confirmed
* non-anemic status (for the control group) based on blood test results
* Resident in the study area for at least 6 months prior to enrollment
* Availability of parental or guardian consent to participate in the study and willingness to follow study protocols
* Completion of all baseline assessments, including neurodevelopmental and physical growth evaluations

Exclusion Criteria:

* Presence of congenital or chronic illnesses that could affect
* neurodevelopment, such as Down syndrome or cerebral palsy.
* History of severe infections or trauma within 3 months prior to enrollment that
* could influence neurodevelopmental outcomes
* Current use of medications or treatments that may interfere with iron metabolism (e.g., iron supplementation or blood transfusions in the last 6 months)
* Premature birth (before 37 weeks of gestation) or low birth weight (< 2,500 grams)
* Parental refusal to provide consent or non-compliance with study procedures.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of children aged 6 to 24 months who attend children health care clinics for routine health check-ups and vaccinations. Participants will be recruited from both hospitals and community health centers within the designated region. The population will include children diagnosed with iron-deficiency anemia and non-anemic controls, providing a comparative sample. The study will aim to capture a diverse range of children from various socioeconomic backgrounds. Informed consent will be obtained from the parents or guardians before participation, and all children will meet the specified inclusion criteria for neurodevelopmental and physical growth evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Development Score | Baseline assessment and follow-up at 6 months.
  This measure assesses neurobehavioral development, including motor skills, language, social behavior, and adaptability, using the "Neuropsychological Behavioral Development Scale for Children Aged 0-6." The score is used to determine the developmental status of children in both the iron-deficiency and non-anemic groups.
Hemoglobin (Hb) | Blood samples will be taken at baseline and follow-up at 3 months.
  To assess the severity of anemia.
Serum Ferritin | Blood samples will be taken at baseline and follow-up at 3 months
  To evaluate the iron stores in the body

SECONDARY OUTCOMES:
Physical Growth (Height) | Baseline assessment and follow-up at 6 months.
  This measure evaluates the physical growth of children, specifically tracking changes in height. Growth data will be compared between children with iron-deficiency anemia and those without to assess the impact of anemia on physical development.
Physical Growth ( Weight) | Baseline assessment and follow-up at 6 months.
  This measure evaluates children's changes in weight. Weight data will be compared between children with and without iron-deficiency anemia to assess anemia's impact on their physical development.
Physical Growth (BMI) | Baseline assessment and follow-up at 6 months.
  This measure assesses children's physical growth by tracking changes in BMI. BMI (Body Mass Index) is calculated by dividing a child's weight (kg) by the square of their height (m²). BMI values will be compared between children with and without iron-deficiency anemia to evaluate anemia's impact on physical development.
Eating behavior | Collected at baseline.
  Eating behavior was assessed using the Children's Eating Behaviour Questionnaire (CEBQ), which evaluates various aspects of children's eating habits, such as food responsiveness, enjoyment of food, and satiety responsiveness. The CEBQ scores will be compared between children with and without iron-deficiency anemia to evaluate how anemia might impact their eating behavior and, in turn, their physical development.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Pingshan District Maternity & Child Healthcare Hospital, Department of Child Healthcare, Shenzhen, China/Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Researchers interested in accessing the individual participant data (IPD) and supporting information can submit a formal request via email to moujs@foxmail.com. Access will be granted to qualified researchers from academic or research institutions, and they will receive de-identified IPD along with supporting documents like the study protocol and statistical analysis plan. Requests must include a research proposal and will be reviewed for compliance with ethical and privacy standards.

REFERENCES:
- [Background] Hanson MA, Gluckman PD. Developmental origins of health and disease--global public health implications. Best Pract Res Clin Obstet Gynaecol. 2015 Jan;29(1):24-31. doi: 10.1016/j.bpobgyn.2014.06.007. Epub 2014 Aug 19. PMID 25225058
- [Background] Pala E, Erguven M, Guven S, Erdogan M, Balta T. Psychomotor development in children with iron deficiency and iron-deficiency anemia. Food Nutr Bull. 2010 Sep;31(3):431-5. doi: 10.1177/156482651003100305. PMID 20973463
- [Background] Georgieff MK. Iron assessment to protect the developing brain. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1588S-1593S. doi: 10.3945/ajcn.117.155846. Epub 2017 Oct 25. PMID 29070550
- [Background] Chikani UN, Bisi-Onyemaechi A, Ohuche I, Onu J, Ugege S, Ogugua C, Mbanefo N, Chime P, Emodi I. The effect of sickle cell anemia on the linear growth of Nigerian children. J Pediatr Endocrinol Metab. 2021 Jul 19;34(10):1283-1290. doi: 10.1515/jpem-2021-0232. Print 2021 Oct 26. PMID 34271599
- [Background] Pivina L, Semenova Y, Dosa MD, Dauletyarova M, Bjorklund G. Iron Deficiency, Cognitive Functions, and Neurobehavioral Disorders in Children. J Mol Neurosci. 2019 May;68(1):1-10. doi: 10.1007/s12031-019-01276-1. Epub 2019 Feb 18. PMID 30778834
- [Background] Yang W, Liu B, Gao R, Snetselaar LG, Strathearn L, Bao W. Association of Anemia with Neurodevelopmental Disorders in a Nationally Representative Sample of US Children. J Pediatr. 2021 Jan;228:183-189.e2. doi: 10.1016/j.jpeds.2020.09.039. Epub 2020 Oct 7. PMID 33035572
- [Background] Stevens GA, Finucane MM, De-Regil LM, Paciorek CJ, Flaxman SR, Branca F, Pena-Rosas JP, Bhutta ZA, Ezzati M; Nutrition Impact Model Study Group (Anaemia). Global, regional, and national trends in haemoglobin concentration and prevalence of total and severe anaemia in children and pregnant and non-pregnant women for 1995-2011: a systematic analysis of population-representative data. Lancet Glob Health. 2013 Jul;1(1):e16-25. doi: 10.1016/S2214-109X(13)70001-9. Epub 2013 Jun 25. PMID 25103581
- See also: The Global Prevalence of Anaemia in 2011 — https://www.who.int/publications/i/item/9789241564960